CLINICAL TRIAL: NCT04601584
Title: Dose-escalation Sequention Cohort Study of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GNR-084 in Patients With Refractory or Relapse Acute Lymphoblastic B-cell Precursor Leukemia.
Brief Title: GNR-084 Safety and Pharmacological Characteristics in Refractory or Relapse B-cell Precursor ALL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BIM-HEM-I; #652 eff date 12.11.2019 (Other: Ministry of Health of Russian Federation)
Record Dates: First submitted 2020-10-13; First posted 2020-10-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: B-precursor Acute Lymphoblastic Leukemia; ALL; GNR-084
Keywords: Leukemia; GNR-084; ALL; Blood Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphoid; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Neoplastic Processes; Pathologic Processes; Antineoplastic Agents
MeSH Terms: conditions — Leukemia; Hematologic Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphoid; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Neoplastic Processes; Pathologic Processes

STUDY DESIGN:
Intervention Model Description: Sequential dose-escalation cohorts in B-ALL patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- GNR-084, dose level 1 (Experimental): Anti-CD19/CD3 antibody
  Interventions: Biological: Cohort 1, GNR-084
- GNR-084, dose level 2 (Experimental): Anti-CD19/CD3 antibody
  Interventions: Biological: Cohort 2, GNR-084
- GNR-084, dose level 3 (Experimental): Anti-CD19/CD3 antibody
  Interventions: Biological: Cohort 3, GNR-084
- GNR-084, dose level 4 (Experimental): Anti-CD19/CD3 antibody
  Interventions: Biological: Cohort 4, GNR-084
- GNR-084, dose level 5 (Experimental): Anti-CD19/CD3 antibody
  Interventions: Biological: Cohort 5, GNR-084
- GNR-084, dose level 6 (Experimental): Anti-CD19/CD3 antibody
  Interventions: Biological: Cohort 6, GNR-084

INTERVENTIONS:
Biological: Cohort 1, GNR-084 — 0.01 ng/kg 6-hours intravenous infusion once a week; 4 doses per cycle, up to 5 cycles
  Other Names: Anti-CD19/CD3 antibody
  Arms: GNR-084, dose level 1
Biological: Cohort 2, GNR-084 — 0.1 ng/kg 6-hours intravenous infusion once a week; 4 doses per cycle, up to 5 cycles
  Other Names: Anti-CD19/CD3 antibody
  Arms: GNR-084, dose level 2
Biological: Cohort 3, GNR-084 — 1 ng/kg 6-hours intravenous infusion once a week; 4 doses per cycle, up to 5 cycles
  Other Names: Anti-CD19/CD3 antibody
  Arms: GNR-084, dose level 3
Biological: Cohort 4, GNR-084 — 4 ng/kg 6-hours intravenous infusion once a week; 4 doses per cycle, up to 5 cycles
  Other Names: Anti-CD19/CD3 antibody
  Arms: GNR-084, dose level 4
Biological: Cohort 5, GNR-084 — 10 ng/kg 6-hours intravenous infusion once a week; 4 doses per cycle, up to 5 cycles
  Other Names: Anti-CD19/CD3 antibody
  Arms: GNR-084, dose level 5
Biological: Cohort 6, GNR-084 — 20 ng/kg 6-hours intravenous infusion once a week; 4 doses per cycle, up to 5 cycles
  Other Names: Anti-CD19/CD3 antibody
  Arms: GNR-084, dose level 6

SUMMARY:
It is an open-label dose-escalating study in sequential cohorts to assess safety and pharmacokinetics of GNR-084.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemias (ALL) are a heterogeneous group of malignant clonal diseases of the blood system originating from precursor cells of hematopoiesis, predominantly of lymphoid differentiation.

More than 7,200 new cases of ALL are diagnosed annually in the European Union (EU), with approximately 40% (approximately 3,000 cases) occurring in adults The main reason for the failure of treatment of acute B-cell lymphoblastic leukemias (B-ALL) is the primary refractoriness to chemical exposure and relapses of the disease, which actually occur in 40-50% of adult patients with ALL. The prognosis in these cases is regarded as extremely unfavorable. Escalation of the chemotherapeutic approach is associated with the development of severe toxic infectious and hemorrhagic complications.

The active substance of the preparation GNR-084 is a bispecific antibody to CD19 / CD3 in the BiMS format (bispecific IgG-like molecules).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed informed consent form to participate in the study;
2. Men and women between aged 18 to 45 inclusive;
3. Patients with incurable morphologically / immunophenotypically confirmed refractory/ relapse of B-cell precursors CD19-positive acute lymphoblastic leukemia from (Ph "-" or Ph "+").
4. Two or more previous lines of anti-leucosis therapy.
5. 5-50% of bone marrow blast cells at screening;
6. Functional status on the scale of the Eastern Cooperative Oncology Group (ECOG) 0-2 points at the screening;
7. Life expectancy ≥ 60 days;

Exclusion Criteria:

1. Hematopoietic stem cells transplantation within 12 weeks prior to study inclusion;
2. Active and widespread chronic graft versus host (GVHD) reaction (grade II-IV), including taking immunosuppressants for the prevention and treatment of GVHD within 2 weeks prior the GNR-084 infusion;
3. Investigator and / or sponsor has doubts that patient will complete the study due to rapid disease progression;
4. Chemotherapeutic agent using within 14 days prior the first GNR-084 infusion;

   Exceptions:
   * Emergency leukapheresis;
   * Emergency hydroxyurea using due to hyperleukocytosis for ≤ 7 days;
   * Other supportive care, including antibiotics, at Investigator's discretion
5. Biochemical blood test:

   * The level of total bilirubin> 1.5 upper limit of norm;
   * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT)> 3 upper limit of norm;
   * Glomerular filtration rate (GFR) level ≤30 (СKD-EPI)
6. Medical history of blinatumomab and other bispecific antibodies using;
7. Persistent toxicity event of 3rd and 4th severity degrees (CTCAE ver 5.0) due to previous treatment;
8. HIV-positive status and / or detection of any hepatitis B and / or hepatitis C blood markers;
9. Severe cardiovascular diseases: uncontrolled arterial hypertension, New York Heart Association (NYHA) functional class III or IV chronic heart failure, unstable angina pectoris, stroke, myocardial infarction, transient ischemic attack, coronary artery bypass grafting and coronary revascularization within last 12 months, or signs of pericardial effusion;
10. Individual sensitivity to:

    * GNR-084 components / excipients;
    * human or humanized investigational drug antibodies;
11. Major surgical interventions, accompanied by hospitalization and anesthesia application within 30 days before the patient is included in the study (biopsy is not a significant surgical intervention);
12. Any other malignant neoplasm presence at the present time or within 5 years prior to inclusion in the study;
13. Known suspected Central Nervous System (CNS) lesion by any genesis now or in medical history, including, but not limited to: neuroleukemia, epilepsy, ischemic or hemorrhagic stroke, severe traumatic brain injury, dementia, Parkinson's disease, organic brain damage, cerebellar disorders, psychosis;
14. Extramedullary lesion of any localization;
15. Other clinical trials participation within 30 days before screening;
16. Mental, physical and other reasons hindering patient to adequately assess their behavior and correctly comply with the conditions of the research protocol;
17. Pregnancy and / or lactation;
18. Male and female patients refusal to use adequate methods of contraception throughout the study;
19. Drug addiction;
20. Alcohol addiction.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
GNR-084 safety and tolerability. | Week 10
  The GNR-084 safety and tolerability will be assessed based on an analysis of the frequency of adverse events (AEs) over the period of treatment and observation of patients

SECONDARY OUTCOMES:
The frequency of specific toxicity events | Week 104
GNR-084 Peak Plasma Concentration (Cmax) | First infusion: 5 minutes before administration, immediately after infusion, 30 minutes, 1, 3, 6, 12, 18, 24, 48, 72, 96 hours after infusion.
GNR-084 area under the plasma concentration versus time curve (AUC) | First infusion: 5 minutes before administration, immediately after infusion, 30 minutes, 1, 3, 6, 12, 18, 24, 48, 72, 96 hours after infusion.
GNR-84 half-life (T1/2) | First infusion: 5 minutes before administration, immediately after infusion, 30 minutes, 1, 3, 6, 12, 18, 24, 48, 72, 96 hours after infusion.
GNR-084 elimination rate constant (Kel) | First infusion: 5 minutes before administration, immediately after infusion, 30 minutes, 1, 3, 6, 12, 18, 24, 48, 72, 96 hours after infusion.
GNR-084 mean retention time (MRT) | First infusion: 5 minutes before administration, immediately after infusion, 30 minutes, 1, 3, 6, 12, 18, 24, 48, 72, 96 hours after infusion.
GNR-084 overall clearance (Cl) | First infusion: 5 minutes before administration, immediately after infusion, 30 minutes, 1, 3, 6, 12, 18, 24, 48, 72, 96 hours after infusion.
GNR-084 kinetic volume of distribution (Vz) | First infusion: 5 minutes before administration, immediately after infusion, 30 minutes, 1, 3, 6, 12, 18, 24, 48, 72, 96 hours after infusion.
Peripheral blood B-lymphocyte depletion (CD19, CD20). | First infusion: 5 minutes before administration, 30 minutes, 1, 24, 48, 96 and 144 hours after infusion. Other infusions: 5 minutes before administration and 1 hour after infusion
CD45+ peripheral cell count | First infusion: 5 minutes before administration, 30 minutes, 1, 24, 48, 96 and 144 hours after infusion. Other infusions: 5 minutes before administration and 1 hour after infusion
Peripheral T-lymphocytes count (CD3, CD4, CD8) | First infusion: 5 minutes before administration, 30 minutes, 1, 24, 48, 96 and 144 hours after infusion. Other infusions: 5 minutes before administration and 1 hour after infusion
Peripheral T-memory cells (CD45RA+, CD28+, CCR7+) count | First infusion: 5 minutes before administration, 30 minutes, 1, 24, 48, 96 and 144 hours after infusion. Other infusions: 5 minutes before administration and 1 hour after infusion
Peripheral B-cells/T-cells ratio | First infusion: 5 minutes before administration, 30 minutes, 1, 24, 48, 96 and 144 hours after infusion. Other infusions: 5 minutes before administration and 1 hour after infusion
Cytokine dynamics | First infusion: 5 minutes before administration, 30 minutes, 1, 24, 48, 96 and 144 hours after infusion. Other infusions: 5 minutes before administration and 1 hour after infusion
Immunogenicity | Week 33
Objective response rate (ORR) | After 2 and 5 GNR-084 cycles (each cycle is 28 days)
Complete clinical and hematological remission rate (CR) | After 2 and 5 GNR-084 cycles (each cycle is 28 days)
Frequency of complete remission with incomplete restoration of blood cellularity (CRi) | After 2 and 5 GNR-084 cycles (each cycle is 28 days)
Duration of an objective response (DoR) | Week 104
Relapse-free survival (RFS) | Week 104
Event-free survival (EFS) | Week 104
Overall survival (OS) | Week 104
Minimal residual disease (MRD) (-) rate in CR-patient | After 5 GNR-084 cycles (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, Study Chair — AO GENERIUM
Locations (3):
- Russia (3):
  - Federal State Budget Funded Institution National Medical Research Center of Hematology, Ministry of Health of the Russian Federation (MoH of Russia), Moscow
  - Almazov National Medical Research Centre, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- See also: Clinical trial registry, Ministry of Health of Russian Federation — https://grls.rosminzdrav.ru/CIPermissionMini.aspx?CIStatementGUID=130bc5af-076e-46a8-b8c4-3391f5688540&CIPermGUID=46966D05-6364-48D8-A949-75E71F78EADC